CLINICAL TRIAL: NCT00869700
Title: Pharmacokinetic Interaction Between the Antimalarial Combination Artemether/Lumefantrine and Combination Antiretroviral Therapy Including Lopinavir/Ritonavir in HIV-infected Adults
Acronym: SEACAT 2_4_2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cape Town (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Professor Karen I Barnes, University of Cape Town
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SEACAT 2_4_2; NHREC
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Last update posted 2010-06-28 (Estimated); Status verified 2010-06

CONDITIONS: HIV Infections; Malaria
Keywords: HIV; Malaria; Pharmacokinetics; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Malaria | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Artemether/Lumefantrine — 80mg artemether/480mg lumefantrine
  Trade name: Coartem
  Indication: for management of non-severe malaria

SUMMARY:
Despite the clinical significance of potential interactions between antimalarials and antiretrovirals, no drug interaction studies have been published and there is an urgent need to address this gap in current knowledge.

The aim of the study is to investigate the pharmacokinetics (PK) of antimalarial combination artemether/lumefantrine (AL) and combination antiretroviral therapy (cART) including lopinavir/ritonavir (LPV/r) in HIV-infected adults.

ELIGIBILITY:
Inclusion Criteria:

* Informed and given ample time and opportunity to think about participation and willing and able to comprehend and comply with all trial requirements. The participant has given written informed consent to participate in the study and to abide by study restrictions.
* Male or female subjects of 18 years of age or older.
* HIV-infected as documented by positive HIV-antibody test and confirmed by Western blot.
* Body weight more than 35kg with a body mass index (BMI) ranging between 18.5 to 30kg/m2 inclusive (See Appendix 15.2).
* Karnofsky score above 70 (See Appendix 15.5).
* CD4 count ≥ 200 cells/mm3
* Patients on LPV/r-based cART at stable doses without significant toxicity for at least 6 weeks at screening.

Exclusion Criteria:

* Patients diagnosed with malaria
* Contraindications to artemether/lumefantrine:
* Hypersensitivity to the artemether, lumefantrine or to any of the excipients of Coartem®.
* Pregnant (as confirmed by an HCG test performed at screening) or breast-feeding female.
* Patients with a family history of congenital prolongation of the QTc interval or sudden death or with any other clinical condition known to prolong the QTc interval such as patients with a history of symptomatic cardiac arrhythmias, with clinically relevant bradycardia or with severe cardiac disease.
* Patients with known disturbances of electrolyte balance e.g. hypokalaemia or hypomagnesaemia.
* Patients taking any drug which is metabolised by the cytochrome enzyme CYP2D6 (e.g. flecainide, metoprolol, imipramine, amitriptyline, clomipramine) or CYP3A4.
* Patients taking drugs that are known to prolong the QTc interval such as antiarrhythmics of classes IA and III, neuroleptics, antidepressive agents, certain antibiotics including some agents of the following classes: macrolides, fluoroquinolones, imidazole, and triazole antifungal agents, certain non-sedating antihistaminics (terfenadine, astemizole), cisapride.
* Haemoglobin below 8.5g/dL for female and 9.5g/dL for male subjects.
* Relevant history or current condition(s) that might interfere with drug absorption, distribution, metabolism or excretion.
* Current smokers, or subjects who have stopped smoking less than 3 months prior to the date of screening.
* History of, or current, substance abuse problem or a positive urine screen for drugs of abuse.
* History of alcohol abuse.
* The subject has consumed any alcohol, grapefruit or caffeine-containing products (ie tea, coffee, cola, chocolate) within 24 hours before any dose of AL during each PK profile.
* The subject has participated in strenuous exercise within 24 hours before any AL dose.
* Severely ill or suffering from any serious underlying disease (particularly cardiac, hepatic or renal disease) that in the opinion of the Investigator would make the participant unsuitable for the study in terms of their safety or study analysis.
* The volunteer has participated in another study with any investigational product within 8 weeks before the first administration of the current investigational products, or until at least 5 x t½ elimination has lapsed, whichever is the greater.
* Subjects who, in the opinion of the Investigator, should not participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-06; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Lumefantrine concentration | day 7

CONTACTS AND LOCATIONS:
Overall Officials: Karen I Barnes, MBChB MMed(clin pharm), Principal Investigator — University of Cape Town
Locations (1):
- Groote Schuur Hospital, Ward J51, Old Main Building, Cape Town, Western Province, South Africa

REFERENCES:
- [Derived] Kredo T, Mauff K, Workman L, Van der Walt JS, Wiesner L, Smith PJ, Maartens G, Cohen K, Barnes KI. The interaction between artemether-lumefantrine and lopinavir/ritonavir-based antiretroviral therapy in HIV-1 infected patients. BMC Infect Dis. 2016 Jan 27;16:30. doi: 10.1186/s12879-016-1345-1. PMID 26818566